CLINICAL TRIAL: NCT04607941
Title: Study of Socio-demographic Factors, Behaviors and Practices Associated With Infection With SARS-CoV-2
Brief Title: Study of Socio-demographic Factors, Behaviors and Practices Associated With Infection With SARS-CoV-2 Responsible for COVID-19
Acronym: ComCor
Status: Completed | Type: Observational
Sponsor: Institut Pasteur (Industry)
Collaborators: National Health Insurance Fund (Other); IPSOS (Industry); Institut de Recherche en Santé Publique, France (Other); Université de Nantes (Other); Assistance Publique - Hôpitaux de Paris (Other); iPLesp (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-047; 2020-A02560-39 (Other: ID-RCB)
Record Dates: First submitted 2020-10-20; First posted 2020-10-29 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2022-04

CONDITIONS: Covid19
Keywords: Covid19; behavior; epidemiology; questionnaires
MeSH Terms: conditions — COVID-19; Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cases: Subjects diagnosed as positive for SARS-CoV-2 infection
  Interventions: Other: Questionnaires; Other: Phone interviews
- Close Subjects: Subjects living within the same household as cases:
  * close cases if tested positive for SARS-CoV-2 following contact tracing recommendations
  * close controls if tested negative for SARS-CoV-2 following contact tracing recommendations
  Interventions: Other: Questionnaires; Other: Phone interviews
- Control Subjects: Controls selected within the population to allow for an age, gender and location of residence-matched analysis with cases
  Interventions: Other: Questionnaires; Other: Phone interviews

INTERVENTIONS:
Other: Questionnaires — Self-administered questionnaires
Other: Phone interviews — A small amount of subjects will be selected at random for phone interviews.

SUMMARY:
The objective of the study is to identify socio-demographic factors, behaviors and practices associated with infection with SARS-CoV-2 to help determine where and how patients mostly get infected with SARS-CoV-2.

It is a case-control study including :

* cases identified by the nationwide system of positive SARS-CoV-2 tests (COVID-19 diagnosis information system, SIDEP) (currently limited to qRT-PCR) and invited to participate by the National Health Insurance (CNAM) which hosts the data from the nationwide test system;
* controls included via Ipsos, a polling institute with access to personal data from a panel from which they will include controls matched on age (divided into 10-year categories), gender and geographic area (departement);
* cases will be offered to invite a person they live with to participate in the study offering another case-control analysis inside a household. These participants will be required to report the result of the test as recommended by contact tracing guidelines to determine whether they are cases or controls.

Data will be collected via a self-administered online questionnaire. Some of the participants will be called for a complementary telephone questionnaire to measure reliability of online retrieved data and explore more specific aspects of SARS-CoV-2 transmission.

DETAILED DESCRIPTION:
The objective of the study is to identify socio-demographic factors, behaviors and practices associated with infection with SARS-CoV-2 to help determine where and how patients mostly get infected with SARS-CoV-2.

The study will focus on sociodemographic data (age, gender, location of residence, socio-economic level, etc.), behaviors and practices (adherence to hand-washing, mask-wearing, work habits, meetings, etc.), the places they visit (public transportation, bars, restaurants, sport facilities, etc.).

It is a case-control study including :

* cases identified by the nationwide system of positive SARS-CoV-2 tests (SIDEP) (currently limited to RT-PCR) and invited to participate by CNAM, which hosts the data from the nationwide test system, through a nationwide email campaign sent once a week; cases will be asked if they can tell where they most probably were infected, leading to a detailed description of the circumstances of the contamination, including whether the suspected contamination took place within the household or not.
* controls included via Ipsos, a polling institute with access to personal data from a panel from which they will include controls matched on age (divided into 10-year categories up to 68 years old included as expected adherence to an online questionnaire quickly drops beyond that age), gender and geographic area (departement); invitations will be sent every week via email to adapt the profile of recruited controls to the age, gender and geographic profiles of the cases that participated in the previous week;
* cases will be offered to invite a person they live with to participate in the study offering another case-control analysis inside a household. Cases will be recommended not to invite the person that they suspect was responsible for their contamination, if a intra-household contamination is suspected. They will indicate the email address of that person to allow sending of an invitation via email. These participants will be required to report the result of the test as recommended by contact tracing guidelines to determine whether they are cases or controls.

Analysis will also include descriptive analysis:

* Estimation of the proportion of cases infected within the household or outside
* Among the cases with a extra-household contamination suspicion, proportion of cases for whom infection circumstances are known and description of these circumstances
* Proportion of cases for whom no specific circumstance of contamination could be evidenced.

Questionnaires will focus on the 10 days preceding :

* symptom onset (symptomatic cases)
* day of testing (asymptomatic cases)
* day of symptom onset of the first case within a household (people from the same household as cases) or testing of the first case if they are asymptomatic
* questionnaire completion (Ipsos-recruited controls)

Participants will be offered at the end of the online self-administered questionnaire to indicate a phone number. Among those agreeing to do so, a random sample of case-control pairs and cases of particular interest (eg with specific contamination circumstances) will be called within two weeks following the online questionnaire for a more detailed telephone questionnaire to measure reliability of online retrieved data and explore more specific aspects of SARS-CoV-2 transmission.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Aged 18 years or more
* Agreeing to participate in the study

Index cases:

* Cases identified by the National Health Insurance (CNAM) in the nationwide database SIDEP (COVID-19 diagnosis information system)
* Positive SARS-CoV-2 RT-PCR on nasopharyngeal or throat swab (or another sample which state of the art considers that it indicates an active infection if positive)

"Distant" controls:

* Selected by Ipsos among Ipsos' panel on age, gender and location of residence criteria (to allow for matched case-control analysis)
* Health Care Workers

Close subjects:

* People who live in the same household as a case and who have been invited to participate by that case
* People who have had a RT-PCR test on nasopharyngeal or throat swab (or another sample which state of the art considers it indicates an active infection if positive) following diagnosis of the index case (following contact tracing recommendations), classified as:
* close cases if test is positive
* close controls if test is negative

Exclusion Criteria:

For all participants:

* People under judicial protection measures ("sauvegarde de justice", "curatelle", "curatelle renforcée", "tutelle", ie various forms of curatorship under French law)

For related cases, related controls and "distant" controls:

* People with a history of SARS-CoV-2 infection confirmed by RT-PCR or positive testing of anti-SARS-CoV-2 antibodies with serology (for related cases: before the current episode)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Index cases: People with positive SARS-CoV-2 test identified by the National Health Insurance (CNAM) in the nationwide database SIDEP (COVID-19 diagnosis information system), which is a system that collects data from tests performed in all testing facilities in France. Only people who have given their e-mail address to the CNAM will be contacted.
  Close subjects: Invited by index cases with whom they live. "Distant" controls: Selected by Ipsos' panel on age, gender and location of residence criteria (to allow for matched case-control analysis) and Health Care Workers.
Sampling Method: Non-Probability Sample
Enrollment: 766818 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Odds-ratios of SARS-CoV-2 infection on socio-demographic factors, behaviors and practices and visited places reported by the participants in the online questionnaire | 1 year
  Odds-ratios of SARS-CoV-2 infection on socio-demographic factors, behaviors and practices and visited places through case-control analyses.

SECONDARY OUTCOMES:
Proportion of cases infected in family environment by SARS-CoV-2 reported by participants in the phone interview | 1 year
  Proportion of cases reporting likely contamination circumstances in the family environment
Proportion of cases infected in family environment by SARS-CoV-2 reported by participants in the online questionnaire | 1 year
  Proportion of cases reporting likely contamination circumstances in the family environment
Proportion of cases infected in professional environment by SARS-CoV-2 reported by participants in the phone interview | 1 year
  Proportion of cases reporting likely contamination circumstances in the professional environment
Proportion of cases infected in professional environment by SARS-CoV-2 reported by participants in the online questionnaire | 1 year
  Proportion of cases reporting likely contamination circumstances in the professional environment
Level of adherence to mask-wearing reported in the phone interview | 1 year
  Proportion of participants reporting adherence to mask-wearing
Level of adherence to mask-wearing reported in the online questionnaire | 1 year
  Proportion of participants reporting adherence to mask-wearing
Level of adherence to hand-washing in the phone interview | 1 year
  Proportion of participants reporting adherence to hand-washing
Level of adherence to hand-washing in the online questionnaire | 1 year
  Proportion of participants reporting adherence to hand-washing
Odds-ratios of SARS-CoV-2 infection on socio-demographic factors, behaviors and practices and visited places reported by the participants in the phone interview | 1 year
  Odds-ratios of SARS-CoV-2 infection on socio-demographic factors, behaviors and practices and visited places through case-control analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Fontanet, Pr, Principal Investigator — Institut Pasteur
Locations (2):
- France (2):
  - Caisse Nationale d'Assurance Maladie, Paris
  - IPSOS, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lievre G, Sicsic J, Galmiche S, Charmet T, Fontanet A, Mueller J. Are psychological attitudes towards vaccination an expression of personality? A cross-sectional study on COVID-19 vaccination in France. BMC Public Health. 2025 Jan 17;25(1):209. doi: 10.1186/s12889-025-21364-9. PMID 39825254
- [Derived] Galmiche S, Charmet T, Rakover A, Cheny O, Omar F, David C, Mailles A, Carrat F, Fontanet A. Risk of SARS-CoV-2 infection in professional settings, shops, shared transport, and leisure activities in France, 2020-2022. BMC Public Health. 2024 Sep 4;24(1):2411. doi: 10.1186/s12889-024-19651-y. PMID 39232732
- [Derived] Lievre G, Sicsic J, Galmiche S, Charmet T, Fontanet A, Mueller JE. Are the 7C psychological antecedents associated with COVID-19 vaccine behaviours beyond intentions? A cross-sectional study on at-least-one-dose and up-to-date vaccination status, and uptake speed among adults in France. Vaccine. 2024 May 22;42(14):3288-3299. doi: 10.1016/j.vaccine.2024.04.024. Epub 2024 Apr 19. PMID 38643038
- [Derived] Rakover A, Galmiche S, Charmet T, Cheny O, Omar F, David C, Martin S, Mailles A, Fontanet A. Source of SARS-CoV-2 infection: results from a series of 584,846 cases in France from October 2020 to August 2022. BMC Public Health. 2024 Jan 30;24(1):325. doi: 10.1186/s12889-024-17772-y. PMID 38287286
- [Derived] Galmiche S, Charmet T, Rakover A, Schaeffer L, Cheny O, von Platen C, Omar F, David C, Mailles A, Carrat F, Fontanet A. Risk of SARS-CoV-2 Infection Among Households With Children in France, 2020-2022. JAMA Netw Open. 2023 Sep 5;6(9):e2334084. doi: 10.1001/jamanetworkopen.2023.34084. PMID 37713194
- [Derived] Galmiche S, Charmet T, Madec Y, Rakover A, Schaeffer L, Cheny O, Omar F, Martin S, Mailles A, Carrat F, Fontanet A. Reduction of SARS-CoV-2 intra-household child-to-parent transmission associated with ventilation: results from a case-control study. BMC Public Health. 2023 Jun 26;23(1):1240. doi: 10.1186/s12889-023-16144-2. PMID 37365557